CLINICAL TRIAL: NCT06895421
Title: A Randomized Controlled Trial of Culturally Adapted Cognitive Behavior Therapy Based Guided Self- Help Manual for Schizophrenia Spectrum Disorder
Brief Title: Culturally Adapted Cognitive Behavior Therapy Based Guided Self-help Manual for Schizophrenia Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Punjab (Other)
Responsible Party: Principal Investigator, Nazish Naureen, Clinical Psychologist Punjab Institute of Mental Health, Lahore, Pakistan, University of the Punjab
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Punjab University PHD thesis
Record Dates: First submitted 2024-08-26; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Receives Treatment As Usual; Receives Culturally Adapted CBTp GSH; Schizophrenia Disorders
Keywords: Schizophrenia Spectrum Disorder, culturally adapted, Guided Self-Help, RCT
MeSH Terms: conditions — Schizophrenia | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: Receives culturally adapted CBTp- GHS plus treatment as usual. (Experimental): Participants receive culturally adapted Cognitive Behaviour Therapy for Psychosis-based Guided Self-Help.
- Group 2: Receives Treatment As Usual (TAU). (Active Comparator): TAU Arm: Participants receive standard treatment as usual.
  Interventions: Drug: Treatment as usual

INTERVENTIONS:
Behavioral: Cognitive behavior therapy based guided self help manual for psychosis plus treatment as usual — The Cognitive Behavior Therapy-Based Guided Self-Help (CBTp-GSH) manual is a structured intervention designed specifically for individuals with psychosis, particularly those diagnosed with Schizophrenia Spectrum Disorders. This manual offers a culturally adapted approach, providing participants with tools and strategies rooted in Cognitive Behavioral Therapy (CBT) principles, tailored to be delivered through guided self-help.
Drug: Treatment as usual — anti psychotic drugs which they are already using
  Arms: Group 2: Receives Treatment As Usual (TAU).

SUMMARY:
The study evaluated the effectiveness of a culturally adapted Cognitive Behaviour Therapy for Psychosis (CBTp) Guided Self-Help (CBTp-GSH) intervention. It involved three phases: a qualitative study for cultural adaptation, a Randomized Controlled Trial (RCT) to test its efficacy against standard treatment, and an assessment of clinician training in applying the intervention. The findings showed that the culturally adapted CBTp-GSH was effective for individuals with Schizophrenia Spectrum Disorder, emphasizing the need for culturally sensitive therapy materials and proper clinician training.

DETAILED DESCRIPTION:
Cognitive Behaviour Therapy for Psychosis (CBTp) is an evidence-based, widely practiced therapy in the Western world. However, it has been underutilized in low and middle-income countries due to the lack of trained therapists and the inadequate cultural adaptation of therapy materials. The study aimed to evaluate the effectiveness of a culturally adapted CBTp-based Guided Self-Help (CBTp-GSH) intervention.

Study I was a qualitative investigation into the cultural adaptation of the CBTp-based Guided Self-Help Manual for individuals with Schizophrenia Spectrum Disorder. The study comprised three phases, which included focus groups, in-depth semi-structured interviews, and panel discussions. Data were analyzed using Thematic Analysis.

Study II involved a Randomized Controlled Trial (RCT) to test the efficacy of the CBTp-GSH Manual for Schizophrenia Spectrum Disorder. A total of 140 patients were equally randomized into two groups: CBTp-GSH or Treatment As Usual (TAU). Assessments were conducted at pre-treatment, post-treatment, and three months post-treatment by blind assessors. The outcome measures included the PANSS, PSYRATS, Insight Scale, and WHO Disability Scale. The results were analyzed using intent-to-treat analysis, incorporating both descriptive and inferential statistics.

Study III focused on the use of Fidelity Assessments to train frontline clinicians in the delivery of the culturally adapted CBTp-based Guided Self-Help Manual. Frontline clinicians were trained and monitored on the application of this intervention in practice cases. The PANSS was utilized to assess psychopathology in clients, and the Revised-Cognitive Therapy for Psychosis Adherence Scale measured therapist fidelity.

The study successfully demonstrated the effectiveness of culturally adapted CBTp-GSH for Schizophrenia Spectrum Disorder and highlighted the importance of training clinicians in delivering culturally sensitive interventions.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria of the present research was

* Clients who could read and write had a minimum of 8th grade education.
* Clients who were able to engage with a mental health professional.
* Both inpatients and outpatients with a diagnosis of Schizophrenia or any Schizophrenia Spectrum Disorder, according to the DSM-V(American Psychiatric Association 2000), was included in the study.
* Client aged 18 to 60 years was included in the research.

Exclusion Criteria:

* Clients with co-morbid conditions such as alcohol or substance dependence, organic
* Brain syndrome, learning disability or high levels of disturbed behavior were excluded from the research. Client with high risk of suicide or homicide based on clinical impression was excluded from the research.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 170 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-05-05 (Actual); Study Completion 2024-08-12 (Actual)

PRIMARY OUTCOMES:
POSITIVE AND NEGATIVE SYMPTOM SCALE | 8 TO 12 WEEKS
  Positive and negative symptom scale was administered on pre and post level to measure the severity of symptoms High score indicates the worse outcome Lower score indicates better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- University of the Punjab, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No